CLINICAL TRIAL: NCT01969175
Title: Effect of a Low-glycemic-load and Milk-free Diet on Acne Severity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Parc Taulí Hospital Universitari (Other)
Responsible Party: Principal Investigator, Lorena Leal, MD, Medical Doctor, Parc Taulí Hospital Universitari
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HPT 2013-059
Record Dates: First submitted 2013-10-21; First posted 2013-10-25 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2013-11

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Diet (Experimental)
  Interventions: Other: Low-glycemic-load and milk-free diet
- Control (Placebo Comparator)

INTERVENTIONS:
Other: Low-glycemic-load and milk-free diet
  Arms: Intervention Diet

SUMMARY:
The objective of this study is to assess the effect of a low-glycemic-load and milk-free diet on acne severity.

IGF-1 and a phosphorylated product of the mTORC pathway (p70S6K) will be assessed in both groups to explore the mTORC signaling pathway, which is thought to be related to clinical improvement in previous studies.

ELIGIBILITY:
Inclusion Criteria:

* Mild, moderate or severe acne (GAGS score 15-44)
* Age: 14-20 years old
* Presence of acne for at least 2 months

Exclusion Criteria:

* Diabetes
* Polycystic ovary syndrome
* Use of hormonal contraceptives
* Previous use of oral retinoids
* Use of oral antibiotics or topical antibacterial or retinoid agents in the last 2 months
* Use of medications known to cause or exacerbate acne including lithium, oral or injected retinoids, some anticonvulsant drugs, medications containing iodides or bromides
* Drug or alcohol abuse.
* Active smokers
* Anticipated difficulty attending visits or fear of blood draws

Ages: 14 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
GAGS Acne severity scale | 13 weeks

SECONDARY OUTCOMES:
Serum insulin like growth factor 1 (IGF-1) | 13 weeks
Diet acceptability and adherence | 13 weeks
p70S6K | 13 weeks
  A phosphorylated product of mTORC signaling pathway

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Parc Taulí, Sabadell, Barcelona, Spain

REFERENCES:
- [Result] Kwon HH, Yoon JY, Hong JS, Jung JY, Park MS, Suh DH. Clinical and histological effect of a low glycaemic load diet in treatment of acne vulgaris in Korean patients: a randomized, controlled trial. Acta Derm Venereol. 2012 May;92(3):241-6. doi: 10.2340/00015555-1346. PMID 22678562
- [Result] Smith RN, Mann NJ, Braue A, Makelainen H, Varigos GA. A low-glycemic-load diet improves symptoms in acne vulgaris patients: a randomized controlled trial. Am J Clin Nutr. 2007 Jul;86(1):107-15. doi: 10.1093/ajcn/86.1.107. PMID 17616769
- [Result] Reynolds RC, Lee S, Choi JY, Atkinson FS, Stockmann KS, Petocz P, Brand-Miller JC. Effect of the glycemic index of carbohydrates on Acne vulgaris. Nutrients. 2010 Oct;2(10):1060-72. doi: 10.3390/nu2101060. Epub 2010 Oct 18. PMID 22253996